CLINICAL TRIAL: NCT00018239
Title: Aging and Cellular Mechanism for Insulin Action After Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: AGCG-001-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise

INTERVENTIONS:
Procedure: Exercise

SUMMARY:
This study will determine whether the metabolic and cellular mechanisms contributing to improved insulin action after aerobic or resistive exercise are different in older, obese, insulin resistant veterans. The hypothesis is that regular exercise, whether aerobic or resistive, will improve whole body insulin action, but the nature and magnitude of changes in skeletal muscle will differ between the two types of exercise.

DETAILED DESCRIPTION:
Veterans will be of comparable body composition and age, and randomly assigned to either aerobic or resistive exercise. They will be instructed in a weight maintenance diet prior to beginning the exercise program, and maintain this diet throughout the study. Metabolic testing will be performed at baseline and after 6 months of exercise training. Testing will include measurement of body composition (anthropometry, dual-energy Xray absorptiometry, computed tomograph scan), maximal oxygen consumption, and muscle strength, glucose tolerance (oral glucose tolerance test), insulin sensitivity (euglycemic-hyperinsulinemic clamp), and muscle biopsies to examine skeletal muscle metabolic characteristics (fiber type distribution, capillary density, oxidative and glycolytic enzyme activities, and levels of key proteins important in insulin signaling and glucose transport). Data will be analyzed using analysis of variance to determine differences between the two exercise groups, and multiple regression analysis to determine the primary adaptations that are associated with the improvements in whole body insulin action.

ELIGIBILITY:
Males between 50 years and 80 years

Overweight

Non-smoker

Sedentary (no regular exercise for one year)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Goldberg, M.D.
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States